CLINICAL TRIAL: NCT05363254
Title: CSD200902: A Study to Assess Indoor Air Quality for a Heated Tobacco Product (20023145 and 20022187) With Four Non-Combusted Cigarette Variants (40007386, 42001399, 42001401, 42001402) in an Environmental Testing Chamber
Brief Title: CSD200902: Assessment of Indoor Air Quality for a Heated Tobacco Product With Four Non-Combusted Cigarette Variants in an Environmental Testing Chamber
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CSD200902
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2022-06

CONDITIONS: Tobacco Use; Smoking; Tobacco Smoking
MeSH Terms: conditions — Tobacco Use; Smoking; Tobacco Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Cohort 1: Marlboro Gold Box (Experimental): Subjects will self-assign to a Cohort 1 based on their self-reported use of Marlboro Gold as their usual brand of combustible cigarettes.
  Interventions: Other: Marlboro Gold Box
- Cohort 2: Newport Box (Experimental): Subjects will self-assign to a Cohort 2 based on their self-reported use of Newport as their usual brand of combustible cigarettes.
  Interventions: Other: Newport Box
- Cohort 3: HTP device with mode A (20023145) and non-combusted cigarette variant 42001401 (Experimental): Subjects will self-assign to one of 6 menthol flavor variant cohorts (Cohort 3 - 8) of non-combusted cigarette products based on their self-reported flavor usage history and a trial use of the 3 menthol flavor variants.
  Interventions: Other: Non-combusted cigarette variant 42001401
- Cohort 4: HTP device with mode B (20022187) and non-combusted cigarette variant 42001401 (Experimental): Subjects will self-assign to one of 6 menthol flavor variant cohorts (Cohort 3 - 8) of non-combusted cigarette products based on their self-reported flavor usage history and a trial use of the 3 menthol flavor variants.
  Interventions: Other: Non-combusted cigarette variant 42001401
- Cohort 5: HTP device with mode A (20023145) and non-combusted cigarette variant 42001399 (Experimental): Subjects will self-assign to one of 6 menthol flavor variant cohorts (Cohort 3 - 8) of non-combusted cigarette products based on their self-reported flavor usage history and a trial use of the 3 menthol flavor variants.
  Interventions: Other: Non-combusted cigarette variant 42001399
- Cohort 6: HTP device with mode B (20022187) and non-combusted cigarette variant 42001399 (Experimental): Subjects will self-assign to one of 6 menthol flavor variant cohorts (Cohort 3 - 8) of non-combusted cigarette products based on their self-reported flavor usage history and a trial use of the 3 menthol flavor variants.
  Interventions: Other: Non-combusted cigarette variant 42001399
- Cohort 7: HTP device with mode A (20023145) and non-combusted cigarette variant 40007386 (Experimental): Subjects will self-assign to one of 6 menthol flavor variant cohorts (Cohort 3 - 8) of non-combusted cigarette products based on their self-reported flavor usage history and a trial use of the 3 menthol flavor variants.
  Interventions: Other: Non-combusted cigarette variant 40007386
- Cohort 8: HTP device with mode B (20022187) and non-combusted cigarette variant 40007386 (Experimental): Subjects will self-assign to one of 6 menthol flavor variant cohorts (Cohort 3 - 8) of non-combusted cigarette products based on their self-reported flavor usage history and a trial use of the 3 menthol flavor variants.
  Interventions: Other: Non-combusted cigarette variant 40007386
- Cohort 9: HTP device with mode A (20023145) and non-combusted cigarette variant 42001402 (Experimental): Subjects will self-assign to one of 2 non-menthol flavor variant cohorts (Cohort 9 and 10) of non-combusted cigarette products based on their self-reported flavor usage history.
  Interventions: Other: Non-combusted cigarette variant 42001402
- Cohort 10: HTP device with mode B (20022187) and non-combusted cigarette variant 42001402 (Experimental): Subjects will self-assign to one of 2 non-menthol flavor variant cohorts (Cohort 9 and 10) of non-combusted cigarette products based on their self-reported flavor usage history.
  Interventions: Other: Non-combusted cigarette variant 42001402

INTERVENTIONS:
Other: Marlboro Gold Box — A combustible cigarette
  Arms: Cohort 1: Marlboro Gold Box
Other: Newport Box — A combustible cigarette
  Arms: Cohort 2: Newport Box
Other: Non-combusted cigarette variant 42001401 — A menthol flavor variant of a non-combusted cigarette (42001401)
  Arms: Cohort 3: HTP device with mode A (20023145) and non-combusted cigarette variant 42001401; Cohort 4: HTP device with mode B (20022187) and non-combusted cigarette variant 42001401
Other: Non-combusted cigarette variant 42001399 — A menthol flavor variant of a non-combusted cigarette (42001399)
  Arms: Cohort 5: HTP device with mode A (20023145) and non-combusted cigarette variant 42001399; Cohort 6: HTP device with mode B (20022187) and non-combusted cigarette variant 42001399
Other: Non-combusted cigarette variant 40007386 — A menthol flavor variant of a non-combusted cigarette (40007386)
  Arms: Cohort 7: HTP device with mode A (20023145) and non-combusted cigarette variant 40007386; Cohort 8: HTP device with mode B (20022187) and non-combusted cigarette variant 40007386
Other: Non-combusted cigarette variant 42001402 — A non-menthol flavor variant of a non-combusted cigarette (42001402)
  Arms: Cohort 10: HTP device with mode B (20022187) and non-combusted cigarette variant 42001402; Cohort 9: HTP device with mode A (20023145) and non-combusted cigarette variant 42001402

SUMMARY:
This is a single-center, open-label, parallel-cohort study to measure and compare the levels of selected secondhand smoke (SHS) constituents of a heated tobacco product (HTP) against combustible cigarettes (CC) after ad libitum smoking sessions by generally healthy smokers in an environmental testing chamber (ETC). Evaluation of SHS constituents detected during non-smoking sessions will be performed as a control.

DETAILED DESCRIPTION:
This study will recruit smokers of both non-menthol and menthol combustible cigarettes, and will allow users of non-menthol and menthol HTPs, and dual users of non-menthol and menthol CCs and HTPs. Safety will be monitored throughout the study by the Principal Investigator (PI) (or designee) by assessing adverse events (AEs), vital sign measurements, standard physical examinations (including oral examinations), electrocardiograms (ECGs), changes in clinical laboratory test results, and pregnancy testing.

Potential subjects will complete a pre-screening telephone interview and a Screening Visit to assess their eligibility within 45 days prior to the Enrollment Visit. The Enrollment visit will occur at least 2 weeks prior to the start of the Chamber Visits. Subjects will be assigned to one of the ten study cohorts based on reported usual brand (UB) CCs and/or HTPs. Cohorts 1 and 2 will use UB CC, Marlboro Gold Box or Newport Box. Subjects in Cohorts 3 through 10 will be assigned to either a non-menthol or menthol HTP investigational products (IP) flavor cohort depending upon past flavor usage history. Subjects will either be assigned to the non-menthol HTP IP or to one of the three menthol HTP IPs after sampling or trying the three menthol HTP IPs and determining which menthol product they would like to use for the length of the study. Once a particular cohort has reached full enrollment, that flavor will no longer be available for sampling and selection. Subjects will be instructed not to use UB CC or HTP during the study.

Subjects assigned to Cohorts 3 through 10 will participate in a 2-week HTP IP familiarization period (prior to Chamber Visit 1), during which subjects will be provided sufficient HTP IP for at-home ad libitum use. The HTP IP includes a battery-powered device, which electronically heats but does not burn tobacco, and requires a non-combusted cigarette, which is inserted into and heated by the HTP device during use. Once heated, the user can begin puffing in the same way as with a CC, on the filter end of the non-combusted cigarette.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an informed consent form (ICF) and complete any questionnaires written in English.
2. Generally healthy male or female adults, 21 years of age or older, inclusive, at the time of signing the ICF.
3. Self-reports at the Screening Visit smoking at least 5 cigarettes per day and inhaling the smoke, for at least 3 months prior to the Screening Visit. Users of HTPs that smoke at least 5 sticks per day will also be allowed into the study. Dual users of combustible cigarettes (CC) and HTPs (either 5 combustible cigarettes or 5 HTP sticks per day, or a combination of 5 CC/HTP products per day) will also be allowed into the study.
4. Positive urine cotinine test at the Screening Visit.
5. Smokes any commercially available brand cigarette as their UB. UB cigarette is defined as the cigarette brand style currently smoked most frequently by the subject. Users of HTPs will also be allowed into the study. Specific brand users must meet the following cohort-specific requirements:

   1. Cohort 1: Self-reports smoking Marlboro Gold Box as their UB and willing to smoke self-provided UB cigarettes for the duration of the study.
   2. Cohort 2: Self-reports smoking Newport Box as their UB and willing to smoke self-provided UB cigarettes for the duration of the study.
   3. Cohorts 3 through 8: Self-reports smoking any style of menthol cigarette as their UB and willing to use a menthol non-combusted cigarette variant ad libitum for the duration of the study. Users of menthol HTPs will also be allowed into this cohort.
   4. Cohorts 9 and 10: Self-reports smoking any style of non-menthol cigarette as their UB and willing to use a non-menthol non-combusted cigarette variant ad libitum for the duration of the study. Users of non-menthol HTPs will also be allowed into this cohort.
   5. For Cohorts 3 through 10: Willing to use the HTP IP during the 2-week at-home ad libitum familiarization period in place of their UB, during the 10 chamber test sessions at the ETC, and at-home during the 2-week period of Chamber Visits in place of their UB.
6. Females must be willing to use a form of contraception acceptable to the Principal Investigator (PI) from the time of signing the ICF until Study Discharge. Examples of acceptable means of birth control are, but not limited to:

   1. Surgical sterilization (hysterectomy, bilateral tubal ligation/occlusion, bilateral oophorectomy, bilateral salpingectomy);
   2. Established use of oral, implantable, injectable, or transdermal methods of contraception associated with inhibition of ovulation;
   3. Physical barrier method (e.g., condom, diaphragm/sponge/cervical cap) with spermicide;
   4. Non-hormone releasing intrauterine devices (IUD) or hormone-releasing IUDs (e.g., Mirena or Kyleena);
   5. Vasectomized partner;
   6. Abstinence from heterosexual intercourse (as a lifestyle choice, not just for the purpose of study participation); and
   7. Post-menopausal and not on hormone replacement therapy.
7. Males must use an acceptable method of birth control from Visit 1 until the end of the study, unless they have had a vasectomy or are abstinent from heterosexual intercourse (as a lifestyle choice, not just for the purpose of study participation), or their female partner is not able to bear children.
8. Able to safely perform the required study procedures, as determined by the PI.

Exclusion Criteria:

1. Presence of clinically significant uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, gastrointestinal, psychiatric, hematological, neurological disease, or any other concurrent disease or medical condition that, in the opinion of the PI, makes the study participant unsuitable to participate in this clinical study.
2. History of, presence of, or clinical laboratory test results indicating diabetes.
3. Systolic blood pressure of > 160 mmHg or a diastolic blood pressure of > 95 mmHg, measured after being seated for five minutes.
4. Scheduled treatment for asthma currently or within the past consecutive 12 months prior to the Screening Visit. As-needed treatment, such as inhalers, may be allowed at the PI's discretion, pending approval from the Medical Monitor.
5. Any history of cancer, except for primary cancers of skin such as localized basal cell/squamous cell carcinoma that have been surgically and/or cryogenically removed.
6. Use of any medication or substance that aids in smoking cessation, including but not limited to any nicotine replacement therapy (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), or lobelia extract within (≤) 30 days prior to the signing of informed consent.
7. Participation in another clinical trial within (≤) 30 days prior to signing the ICF. The 30-day window for each subject will be derived from the date of the last study event in the previous study to the time of signing the ICF in the current study.
8. Females who have a positive pregnancy test, or who are pregnant, are breastfeeding, or intend to become pregnant during the course of the study.
9. Subjects ≥ 35 years of age currently using systemic, estrogen-containing contraception or hormone replacement therapy.
10. A positive urine drug screen without evidence of prescribed corresponding concomitant medication(s) at the Screening Visit or Enrollment Visit, with the exception of for tetrahydrocannabinol (THC). If positive for THC, a cannabis intoxication evaluation will be performed at check-in, and inclusion will be at the discretion of the PI or appropriately qualified designee.
11. Postpones a decision to quit using tobacco- or nicotine-containing products in order to participate in this study or a previous attempt within (≤) 30 days prior to signing the ICF.
12. Drinks more than 21 servings of alcoholic beverages per week or has a positive alcohol test result at the Screening Visit or Enrollment Visit.
13. Employed by a tobacco or nicotine manufacturing company, the study site, or handles tobacco- or nicotine-containing products as part of their job.
14. Regularly exposed to solvent fumes or gasoline (e.g., painter, gas-station mini-mart employee).
15. History of clinically significant claustrophobia.
16. Determined by the PI to be inappropriate for this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Real-time and time-weighted average (TWA) concentrations of Acetaldehyde | 20 minutes
  To assess differences in levels of selected Secondhand smoke (SHS) constituents after ad libitum human use of each non-combusted cigarette variant heated by the HTP device in an environmental testing chamber compared to after ad libitum human smoking of combustible cigarettes
Real-time and time-weighted average (TWA) concentrations of Ammonia (NH3) | 20 minutes
  To assess differences in levels of selected Secondhand smoke (SHS) constituents after ad libitum human use of each non-combusted cigarette variant heated by the HTP device in an environmental testing chamber compared to after ad libitum human smoking of combustible cigarettes
Real-time and time-weighted average (TWA) concentrations of Benzene | 20 minutes
  To assess differences in levels of selected Secondhand smoke (SHS) constituents after ad libitum human use of each non-combusted cigarette variant heated by the HTP device in an environmental testing chamber compared to after ad libitum human smoking of combustible cigarettes
Real-time and time-weighted average (TWA) concentrations of Carbon monoxide (CO) | 20 minutes
  To assess differences in levels of selected Secondhand smoke (SHS) constituents after ad libitum human use of each non-combusted cigarette variant heated by the HTP device in an environmental testing chamber compared to after ad libitum human smoking of combustible cigarettes
Real-time and time-weighted average (TWA) concentrations of Formaldehyde | 20 minutes
  To assess differences in levels of selected Secondhand smoke (SHS) constituents after ad libitum human use of each non-combusted cigarette variant heated by the HTP device in an environmental testing chamber compared to after ad libitum human smoking of combustible cigarettes
Real-time and time-weighted average (TWA) concentrations of Nicotine | 20 minutes
  To assess differences in levels of selected Secondhand smoke (SHS) constituents after ad libitum human use of each non-combusted cigarette variant heated by the HTP device in an environmental testing chamber compared to after ad libitum human smoking of combustible cigarettes
Real-time and time-weighted average (TWA) concentrations of Toluene | 20 minutes
  To assess differences in levels of selected Secondhand smoke (SHS) constituents after ad libitum human use of each non-combusted cigarette variant heated by the HTP device in an environmental testing chamber compared to after ad libitum human smoking of combustible cigarettes
Real-time and time-weighted average (TWA) concentrations of Respirable suspended particulates (RSP) (PM2.5) | 20 minutes
  To assess differences in levels of selected Secondhand smoke (SHS) constituents after ad libitum human use of each non-combusted cigarette variant heated by the HTP device in an environmental testing chamber compared to after ad libitum human smoking of combustible cigarettes

CONTACTS AND LOCATIONS:
Overall Officials: Gary Dull, PhD, Study Director — RAIS
Locations (1):
- Clinical Research Atlanta, Stockbridge, Georgia, United States

IPD SHARING:
Plan to Share IPD: No